CLINICAL TRIAL: NCT04457986
Title: Randomized Controlled Comparison of the Erector Spina Plane Block and Modified Thoracolumbar Interfacial Plane Block and Intravenous Patient Controlled Analgesia in Patients Undergoing Lumbar Disc Surgery
Brief Title: Plane Block vs Intravenous Patient Controlled Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Assoc Professor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESP-MTIP-IVPCA
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-06

CONDITIONS: Lumbar Disc Herniation
Keywords: postoperative pain; erector spina plane block; thoracolumbar interfacial plane block; patient controlled analgesia
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Postoperative pain will be assessed by an anaesthesiologist unaware of group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spina plane block (ESP) (Experimental): Patients will receive Erector spina plane block (ESP) with bupivacaine for postoperative analgesia
  Interventions: Drug: Erector spina plane block (ESP)
- Modified thoracolumbar interfacial plane block (MTI) (Experimental): Patients will receive Modified thoracolumbar interfacial plane block (MTI) with bupivacaine for postoperative analgesia
  Interventions: Drug: Modified thoracolumbar interfacial plane block (MTI)
- Intravenous patient controlled analgesia (IV-PCA) (Active Comparator): Patients will receive Intravenous patient controlled analgesia (IV-PCA) with tramadol for postoperative analgesia
  Interventions: Drug: Intravenous patient controlled analgesia (IV-PCA)

INTERVENTIONS:
Drug: Erector spina plane block (ESP) — Patient will receive ultrasound guided regional anesthesia with bupivacaine and intravenous patient controlled analgesia with tramadol
  Arms: Erector spina plane block (ESP)
Drug: Modified thoracolumbar interfacial plane block (MTI) — Patient will receive ultrasound guided regional anesthesia with bupivacaine and intravenous patient controlled analgesia with tramadol
  Arms: Modified thoracolumbar interfacial plane block (MTI)
Drug: Intravenous patient controlled analgesia (IV-PCA) — Patient will receive intravenous patient controlled analgesia with tramadol
  Arms: Intravenous patient controlled analgesia (IV-PCA)

SUMMARY:
Acute postoperative pain begins with surgical trauma and decreases with tissue healing. Untreatable postoperative pain is one of the most important problems due to the increase in respiratory, cardiac and thromboembolic complications. Lumber disc surgery is widely performed, and patients often complain of postoperative pain.

Preventing and managing postoperative pain after lumber disc surgery is very important for anesthetists. For this purpose, non-steroidal anti-inflammatory agents, intravenous opioids, preemptive analgesia methods, intravenous patient controlled analgesia methods and regional anesthesia techniques are used within the multimodal analgesia strategy.

Regional anesthesia techniques are becoming increasingly widespread due to their efficiency and increased applicability thanks to the use of ultrasonography. Regional anesthesia techniques used in lumber disc surgery include paravertebral block, local anesthetic infiltration, epidural analgesia, and erector spina plan block and modified thoracolumbar interfacial plan block in recent years.

The erector spina plane block was first described in 2016, and the thoracolumbar interfacial plane block in 2015, and its modification was developed in 2017. Although they vary depending on the level of application, they offer analgesic activity in a wide range. Although there are publications about the use of these blocks for postoperative analgesia after lumber surgeries, which block is more effective has not been investigated.

This study may contribute to the development of new options for pain management after lumber disc surgery by comparing erector spina plane block and modified thoracolumbar interfacial plane block, which have recently been used for postoperative pain treatment, with limited research, with each other and the standard technique, intravenous patient controlled analgesia, can add new applications to multimodal analgesia methods, increase patient satisfaction and contribute to the early recovery process.

The objective is to compare the erector spina plane block and modified thoracolumbar interfacial plane block in patients undergoing lumber disc surgery with intravenous patient-controlled analgesia in terms of analgesic efficacy.

Hypothesis The erector spina plane block and modified thoracolumbar interfacial plane block may decrease the postoperative pain scores, opioid consumption and time to first analgesic requirement compared with intravenous patient controlled analgesia.

DETAILED DESCRIPTION:
Patients undergoing lumber disc surgery will be randomised into 3 groups. To receive either Erector spina plane block (ESP) or Modified thoracolumbar interfacial plane block (MTI) or Intravenous patient controlled analgesia IV-PCA.

Patients in the ESP and MTI groups will receive the blocks before anesthesia induction in the preoperative holding area.

All patients will receive IV-PCA with tramadol. Postoperative analgesia will be evaluated with a numeric rating scale at postoperative recovery room admittance, postoperative 1st , second, 4th, 12th and 24th hours both at rest and during movement.

Postoperative tramadol consumption and time to first tramadol demand will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective lumber discectomy or laminectomy
* Adults
* Aged 18-65
* America Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* Emergency surgery
* Chronic pain condition
* Allergic to study drugs
* Recurrent surgical cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Pain score | 10 minutes after extubation
  Pain will be evaluated with the Numeric Rating Scale (0-10 points; 0=no pain and 10=worst pain)
Pain score | postoperative 1st hour
  Pain will be evaluated with the Numeric Rating Scale (0-10 points; 0=no pain and 10=worst pain)
Pain score | postoperative 2nd hour
  Pain will be evaluated with the Numeric Rating Scale (0-10 points; 0=no pain and 10=worst pain)
Pain score | postoperative 4th hour
  Pain will be evaluated with the Numeric Rating Scale (0-10 points; 0=no pain and 10=worst pain)
Pain score | postoperative 12th hour
  Pain will be evaluated with the Numeric Rating Scale (0-10 points; 0=no pain and 10=worst pain)
Pain score | postoperative 24th hour
  Pain will be evaluated with the Numeric Rating Scale (0-10 points; 0=no pain and 10=worst pain)
Tramadol consumption | postoperative 24th hour
  Tramadol consumption will be determined from the ambulatory infusion pump (Abott)
Time to first analgesia request | 10 minutes after extubation
  Time to first tramadol request will be determined from the ambulatory infusion pump (Abott)

CONTACTS AND LOCATIONS:
Overall Officials: ÜNAL Dr YAZICIOĞLU, Assoc Prof, Principal Investigator — DISKAPI YILDIRIM BEYAZIT TEACHING HOSPITAL
Locations (1):
- Ankara Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Result] Ueshima H, Hara E, Otake H. RETRACTED: Thoracolumbar interfascial plane block provides effective perioperative pain relief for patients undergoing lumbar spinal surgery; a prospective, randomized and double blinded trial. J Clin Anesth. 2019 Dec;58:12-17. doi: 10.1016/j.jclinane.2019.04.026. Epub 2019 Apr 25. PMID 31029989 (Retraction: PMID 35393187 J Clin Anesth. 2022 Aug;79:110690)